CLINICAL TRIAL: NCT00327275
Title: The Strength Training and Remicade Study
Brief Title: The Effects of a 16-Week Individualized, Intensive Strength Training Program in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 080192
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2006-05-18 (Estimated); Status verified 2006-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Resistance Training

INTERVENTIONS:
Behavioral: strength training

SUMMARY:
To assess the effects of a 16-week individualized, intensive strength training program in patients with rheumatoid arthritis. Primary and secondary outcomes include: strength and body composition, function, disease activity, pain, quality of life.

We hypothesized that improvements would be seen in all of the above outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with RA
* Over 18 years of age
* ACR Functional Class I and II
* Taking Remicade >4 months

Exclusion Criteria:

* Presence of comorbid conditions contraindicated to exercise, including, but not limited to:

  1. heart disease
  2. severe osteoporosis: (if >50 years): T score < -3.0 for hip or spine excluded; T score <-2.5 for hip or spine w/o current treatment)
  3. (all potential subjects) previous non-traumatic fractures
  4. uncontrolled BP
* BMI >40
* Regular use of assistive walking device which would interfere with ability to lift weights
* Currently or within the last 3 months participating in aerobic exercise > 150 minutes a week
* Currently or within the last 3 months participating in any regular strength training activities
* Presence of neurological impairment that directly limits ability to perform exercise
* Participation in concurrent exercise study
* Any reason for which the investigator deems it would not be in the patient's best interest to continue in the study
* Plans to move away from site within next 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2004-03; Study Completion 2005-01

PRIMARY OUTCOMES:
Strength
Body Composition
Function
Pain

SECONDARY OUTCOMES:
Quality of Life
Disease Activity
Fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Hilary G Flint-Wagner, PhD, MPH, Principal Investigator — Idaho State University
Locations (1):
- University of Arizona, Tucson, Arizona, United States